CLINICAL TRIAL: NCT02922426
Title: A Randomized, Double-Blind, Parallel-Group Study in Healthy Subjects to Characterize Insulin Sensitivity and Lipid Metabolism in Response to Treatment With ALKS 3831 and Olanzapine
Brief Title: An Insulin Sensitivity Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK3831-A108
Record Dates: First submitted 2016-09-30; First posted 2016-10-04 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Healthy Volunteers
Keywords: ALKS 3831; Samidorphan; Olanzapine
MeSH Terms: interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ALKS 3831 (Experimental): Oral, bilayer tablet
  Interventions: Drug: ALKS 3831
- Olanzapine (Active Comparator): Oral, bilayer tablet
  Interventions: Drug: Olanzapine
- Placebo (Placebo Comparator): Oral, bilayer tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALKS 3831 — Daily dosing for 21 consecutive days
  Arms: ALKS 3831
Drug: Olanzapine — Daily dosing for 21 consecutive days
  Arms: Olanzapine
Drug: Placebo — Daily dosing for 21 consecutive days
  Arms: Placebo

SUMMARY:
This study will characterize insulin sensitivity in response to treatment with ALKS 3831, olanzapine, and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18.0 and < 25.0 kg/m^2 at screening and randomization
* No prior history of regular smoking or nicotine use
* Women of child-bearing potential should be on stable regimens of oral contraceptives for at least 2 months prior to screening
* Subjects must be willing to avoid a regular exercise regimen from screening through the end of the treatment period
* Additional criteria may apply

Exclusion Criteria:

* Has current evidence or history of any clinically significant medical or psychiatric condition or observed abnormality
* Is currently pregnant or breastfeeding, or is planning to become pregnant during the study
* Has a lifetime history of diabetes
* Has a known risk of narrow-angle glaucoma
* Has a clinically significant illness within 30 days prior to screening or admission to the clinic
* Has a history of dependence on any substance other than caffeine
* Has a current or anticipated need for prescribed opioid medication (eg, planned surgery) during the study period
* Has a positive urine drug screen for drugs of abuse at screening or admission to the study site
* Has had a serious infection (eg, pneumonia or septicemia) within the 3 months prior to screening or admission to the clinic
* Has had any vaccinations in the 4 weeks prior to screening or admission to the clinic
* Chronic use of non-steroid anti-inflammatory drugs (NSAIDs) and acetaminophen, except for low-dose Aspirin is not allowed
* Use of new prescription and non-prescription drugs, as well as dietary/nutritional supplements within 3 weeks preceding the first dosing of study drugs, unless approved by Investigator
* Has prior use of any antipsychotic medication, including on and off label uses
* Additional criteria may apply

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09; Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Changes in blood glucose concentrations | 21 days
  Differences will be compared among treatment groups

SECONDARY OUTCOMES:
Changes in insulin concentrations | 21 days
  Differences will be compared among treatment groups
Incidence of treatment-emergent adverse events (AEs) | 24 days

CONTACTS AND LOCATIONS:
Overall Officials: David McDonnell, MD, Study Director — Alkermes, Inc.
Locations (1):
- Alkermes Investigational Site, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: Undecided